CLINICAL TRIAL: NCT01170000
Title: Timely End-of-Life Communication to Parents of Children With Brain Tumors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Foundation for Barnes-Jewish Hospital (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Verna Ferguson - Principal Investigator, Barnes-Jewish Hospital
Organization: Barnes-Jewish Hospital (Other)
Other Study IDs: 09-0763 BJH; R21NR011071 (NIH)
Record Dates: First submitted 2010-07-26; First posted 2010-07-27 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Palliative Care; Communication
MeSH Terms: conditions — Communication

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A national priority for health care providers is to initiate early communication about palliative and end-of-life care (PC/EOL) for children with a poor prognosis. Communication about prognosis and advanced care planning is critical to empowering parents to make decisions about PC/EOL for their children. A single-group study to refine and pilot test a PC/EOL communication intervention is entitled, Communication Plan: Early through End of Life (COMPLETE). COMPLETE is designed to be delivered during parent meetings and features: (a) a physician-nurse (MD/RN) team approach to PC/EOL communication; (b) printed visual aids and parent resource forms; and (c) hope and non-abandonment messages tailored by a MD/RN team to their communication style and parental preferences for information. During Phase I, an interdisciplinary approach involving nurses, physicians, PC/EOL expert consultants, and bereaved-parent consultants met to develop a standardized protocol and training procedures. During Phase II, this protocol will be evaluated with 24 parents and MD/RN teams. The investigators will evaluate parental outcomes regarding the COMPLETE's influence on: (a) information needs, emotional needs/resources, appraisal of MD/RN information and of symptom management; and (b) parental distress, uncertainty, decision regret, hope, satisfaction with MD/RN communication, and advance care planning over time. Findings from this study address NIH priorities related to: 1) an underserved population (i.e., parents of children with brain tumors); 2) an under-examined ethical concern about early integration of PC/EOL communication for parents of children with poor prognosis; 3) improved communication about PC/EOL among physicians, nurses, and parents; and 4) the potential for changing health care practice.

DETAILED DESCRIPTION:
Physicians and nurses (MDs/ RNs) struggle to communicate effectively about palliative and end-of-life (PC/EOL) care with parents when their child's prognosis is poor, and rarely collaborate as a team in this difficult process. The aim of this study was to develop and evaluate training strategies for MD/RN dyads to collaboratively deliver a PC/EOL communication intervention called, Communication Plan: Early through End of Life (COMPLETE), to 24 parents of children with brain tumors. During Phase I, training strategies were based on principles from a Relationship Centered Care perspective. The training was delivered to 3 pediatric neuro-oncologists and 5 oncology nurses by a team of parent advisors and a team of expert consultants (i.e., medical ethics, communication, and PC/EOL). Our 2-day training included 4 modules: family assessment, goal directed treatment planning, anticipatory guidance, and staff communication and follow-up. Each module included: didactic content, small group reflective sessions, and communication skills practice with bereaved parent. Evaluations included dichotomous (agree/disagree) ratings and qualitative comments on didactic content, small group reflection, and skills practice for each module. Helpful aspects of our training strategies included: parent advisers' insights, emotional presence, emphasis on hope and non-abandonment messages, written materials to facilitate PC/EOL communication, and a team approach. For this presentation we will discuss insights gained regarding use of a parent advisory panel, strategies to help the MD/RN dyads feel comfortable working as a team to communicate with parents, and ways to improve training procedures and our intervention.

Pediatric oncology physicians and nurses found PC/EOL care communication training strategies and content as helpful and useful. During Phase II of our study, our PC/EOL care communication intervention is planned to be implemented and evaluated with 24 enrolled parents. If effective, this intervention will facilitate integration of quality PC care practices into the care of children with brain tumors.

ELIGIBILITY:
Inclusion Criteria:

* Eligibility criteria include parents who are:
* 18 years of age or older;
* the primary decision makers (i.e., single parent or couple-dyad) for their child (birth to 18 years of age);
* the biological parents, step-parents, or legal guardians (e.g., adoptive parent);
* single or married;
* informed that their child is diagnosed with a brain tumor with a poor prognosis as determined by the primary neuro-oncologist (e.g., glioblastoma multiforme, PNET, WHO grade 3/4 brain tumor, or metastatic medulloblastoma); [3, 33, 38, 41, 42, 175]
* able to read, speak, and understand English.
* Our rationale for these criteria is to include: (a) parents of children who are at high risk of not receiving timely PC/EOL and b) parents who are likely to be mature enough to make difficult decisions on their own. In addition, we recognize the importance of providing sensitive PC/EOL communication to all parents; however, it is beyond the scope of the R21 mechanism to develop scripts in other languages.

Exclusion Criteria:

* Parents will be excluded from the study if:
* the child's brain tumor has a good prognosis (e.g., a non-metastatic medulloblastoma);
* the child has been treated previously for another type of cancer;
* the parents have neurological and/or cognitive impairments, as reported by the site MD/RN team, preventing them from understanding the treatment options and completing the questionnaires;
* either parent in a decision-making couple (i.e., dyad) declines consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The target sample size is 24 parents of 12 children diagnosed with a brain tumor. Our sample size is sufficient to complete descriptive analyses of Aims 2 and 3, and adequate precision for the estimation of effect sizes and preliminary tests of single-arm efficacy in Aim 4.1. This study is powered for adequate estimation of effect sizes, not for efficacy; that is, the study is powered to appropriately detect large effect sizes with lower power for medium effect sizes. If 10% or fewer participants withdraw after COMPLETE Session 1, we will be able to collect data from about 22 parents at least once. Twenty-two parents will provide 61% power for detecting a difference of 0.5 times standard deviation for a two-sided paired t-test with alpha of .05. The same test would have 70% power to detect a difference of .55 standard deviation. This approach is typical and justifiable in pilot feasibility studies to achieve 80% power for detecting only large effect sizes.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Estimated)
Dates: Start 2009-09; Primary Completion 2012-08 (Estimated); Study Completion 2012-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Verna Ferguson, PhD, Principal Investigator — Barnes-Jewish Hospital; Joan Haase, PhD, Principal Investigator — Indiana University
Locations (4):
- United States (4):
  - Riley Children's Hospital, Indianapolis, Indiana
  - Indiana University School of Nursing, Indianapolis, Indiana
  - SSM Cardinal Glennon Children's Hospital, St Louis, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri